CLINICAL TRIAL: NCT01940679
Title: Bioavailability of Encapsulated Omega-3 Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: Combat Feeding Directorate at Natick Soldier, Research, Development and Engineering Center (Unknown)
Responsible Party: Principal Investigator, Tracey Smith, Research Dietitian, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 13-13-H
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Bioavailability of Omega-3s in Military Rations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fresh meat stick (Experimental): Fresh meat stick w/ encapsulated 600 mg EPA/DHA; product frozen immediately after production.
  Interventions: Dietary Supplement: encapsulated 600 mg EPA/DHA
- Stored meat stick (Experimental): Stored meat stick with encapsulated 600 mg EPA/DHA; stored at 100F for 3 months after production
  Interventions: Dietary Supplement: encapsulated 600 mg EPA/DHA
- Fresh pound cake (Experimental): Fresh pound cake w/ encapsulated 600 mg EPA/DHA; product frozen immediately after production.
  Interventions: Dietary Supplement: encapsulated 600 mg EPA/DHA
- Stored pound cake (Experimental): Stored pound cake with encapsulated 600 mg EPA/DHA; stored at 100F for 3 months after production.
  Interventions: Dietary Supplement: encapsulated 600 mg EPA/DHA

INTERVENTIONS:
Dietary Supplement: encapsulated 600 mg EPA/DHA — encapsulated 600 mg EPA/DHA

SUMMARY:
Omega-3 fatty acids (n-3s), particularly eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), have anti-inflammatory properties and other documented beneficial health effects that could warrant n-3 fortification of combat rations. However, military combat rations must meet rigorous shelf-stability guidelines (e.g.,, 3 years at 80°F or 6 months at 100°F), which is problematic for natural food sources of n-3s (e.g., oil and fish), which degrade when exposed to high temperatures and prolonged shelf-storage. Encapsulation, e.g., coating freeze dried n-3s with gelatin, can prevent this degradation, and Natick Soldier Research, Development and Engineering Center's (NSRDEC) Combat Feeding Directorate used encapsulated n-3 technology to produce n-3 enriched ration items that withstand environmental stressors and meet shelf-life specifications for military rations. However, the bioavailability of the encapsulated n-3s in these rations is unknown, particularly when they are incorporated into high-protein food items and exposed to high temperatures and prolonged storage. In this randomized, cross-over study, civilian and/or military personnel will be asked to consume: 1) a high protein food item enriched with encapsulated n-3s (600 mg) and previously stored for 6 months at 100°F; 2) a low-protein food item enriched with encapsulated n-3s (600 mg) and previously stored for 6 months at 100°F; 3) a high protein food item with encapsulated n-3s (600 mg) that was not subjected to high-temperature and prolonged storage; and, 4) a low-protein food item with encapsulated n-3s (600 mg) that was not subjected to high temperature and prolonged storage. Serial blood sampling to measure acute changes in the circulating fatty acid profile will occur in the hour before and 6 hours after consumption of each ration component. The only known risks, which this study presents to participants, are those associated with venous catheter placement. The results will help military ration developers determine the ration components best suited for n-3 fortification.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 45 years old
* leave status and have approval from your supervisor (for DoD Civilians)

Exclusion Criteria:

* under the age of 18 or over the age of 45
* bleeding disorder (von Willebrand disease, hemophilia) or taking medications that impair ability to stop bleeding (heparin)
* consumed ≥1 serving (equivalent to a deck of cards) of salmon, herring, mackerel, anchovies, sardines, halibut or tuna or omega-3 enriched eggs per week over the previous past month
* regularly consume dietary supplements (for example, capsules) containing omega-3 fatty acids

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Plasma n-3 concentrations | 15 minute, 2 hrs, 4 hrs and 6 hrs after consumption of n-3 rich food item

CONTACTS AND LOCATIONS:
Overall Officials: Tracey J Smith, PhD, Principal Investigator — U.S. Army Research Institute of Environmental Medicine
Locations (1):
- U.S. Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States